CLINICAL TRIAL: NCT07250620
Title: Diagnostic Accuracy of 10-Minute Vs 30-Minute CTG in Intrapartum Fetal Monitoring.
Brief Title: Comparison Between Using 10min CTG in Fetal Monitoring Instead of 30min Monitoring in Low Resources Overcrowded Hospitals.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Soliman Mohamed Soliman Alazhary, Dr.Soliman Mohamed Alazhary, Assiut University
Other Study IDs: 10min CTG monitoring accuracy.
Record Dates: First submitted 2025-11-16; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Normal Pregnancy; Labor Active Dilated Cm
Keywords: CTG; Fetal monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- women full term pregenancy in active stage of labor

SUMMARY:
Cardiotocography (CTG) is a cornerstone of intrapartum fetal monitoring but requires a minimum of 30 minutes for a reliable trace, creating a significant bottleneck in high-volume, low-resource settings like Egypt As it is time-consuming and resource intensive. This leads to delays in care and increased workload for healthcare providers. A shortened, yet accurate, CTG protocol could drastically improve workflow and resource allocation without compromising fetal safety.

DETAILED DESCRIPTION:
In Egypt, labor wards in tertiary hospitals are often overcrowded with limited CTG machines and midwives. The requirement of a minimum 30-minute CTG trace creates bottlenecks in care and increases staff workload. Previous studies suggest that the first 10 minutes of a CTG may capture the essential features of fetal well-being. If validated, a shortened CTG could improve efficiency in high-volume maternity units without compromising neonatal outcomes. Using umbilical venous pH as the gold standard for fetal acid-base status, this study will directly compare the diagnostic accuracy of a 10-minute versus a 30-minute CTG protocol in low-risk laboring women. The aim is to evaluate whether a 10-minute CTG tracing is non-inferior to the standard 30 minute CTG in fetal assessment and predicting fetal acid-base status (umbilical venous pH) in term, low-risk pregnancies during the active first stage of labor.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy.
* Gestational age ≥ 37 weeks.
* Vertex presentation.
* Active first stage of labor (cervical dilation ≥ 4 cm).
* Low-risk pregnancy (no hypertension, diabetes, IUGR, or other significant complications).

Exclusion Criteria:

* • Multiple gestation.

  * Known major fetal anomaly.
  * Non-vertex presentation.
  * Indication for continuous CTG (e.g., meconium-stained liquor, antepartum hemorrhage).
  * Maternal refusal.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women only with full term pregnancy
Study Population: All women who come to Women's Health Assiut university hospital in labor and meet the inclusion criteria after informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-17 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To compare the diagnostic accuracy (sensitivity, specificity, PPV, NPV) of a 10 minute CTG versus a standard 30-minute CTG in fetal monitoring and well being | Immediately after birth
  Using fetal acidemia defined as (umbilical venous pH < 7.25) as reference in detecting fetal will being and comparing results with 10-min & 30-min CTG monitoring to evaluate diagnostic accuracy of both in detecting fetal acidemia.

CONTACTS AND LOCATIONS:
Overall Officials: Elwani Eldremey Elsenousy, Professor, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Tomich MF, Leoni RS, Meireles PT, Petrini CG, Araujo Junior E, Peixoto AB. Accuracy of intrapartum cardiotocography in identifying fetal acidemia by umbilical cord blood analysis in low-risk pregnancies. Rev Assoc Med Bras (1992). 2023 May 15;69(6):e20221182. doi: 10.1590/1806-9282.20221182. eCollection 2023. PMID 37194903
- [Result] Alfirevic Z, Devane D, Gyte GM, Cuthbert A. Continuous cardiotocography (CTG) as a form of electronic fetal monitoring (EFM) for fetal assessment during labour. Cochrane Database Syst Rev. 2017 Feb 3;2(2):CD006066. doi: 10.1002/14651858.CD006066.pub3. PMID 28157275
- [Result] Garabedian C, De Jonckheere J, Butruille L, Deruelle P, Storme L, Houfflin-Debarge V. Understanding fetal physiology and second line monitoring during labor. J Gynecol Obstet Hum Reprod. 2017 Feb;46(2):113-117. doi: 10.1016/j.jogoh.2016.11.005. Epub 2017 Jan 30. PMID 28403965
- See also: Related Info — https://www.nice.org.uk/guidance/ng229